CLINICAL TRIAL: NCT01998412
Title: An Open Label, Registry Study of the Safety of Iluvien® 190 Micrograms Intravitreal Implant in Applicator
Brief Title: Iluvien Registry Safety Study
Acronym: IRISS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Alimera Sciences (Industry)
Responsible Party: Sponsor
Organization: ANI Pharmaceuticals (Industry)
Other Study IDs: M-01-12-001
Record Dates: First submitted 2013-11-20; First posted 2013-11-28 (Estimated); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Chronic Diabetic Macular Oedema Considered Insufficiently Responsive to Available Therapies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The study will include any patient treated with Iluvien at designated sites in European countries where marketing authorization has been granted in order to obtain broader safety and usage information.

ELIGIBILITY:
Inclusion Criteria:

* Any patient treated with Iluvien under this protocol will be included in the study.

Exclusion Criteria:

* Patients/Guardians who are unable to understand and sign the Informed Consent will be excluded from the study.

Retrospective Enrollment Criteria

Patients treated with ILUVIEN prior to study initiation may be included provided they satisfy the inclusion and exclusion criteria, where applicable, as well as, the following requirements:

1. The site is allowed to enroll a patient who was treated with ILUVIEN no more than 36 months prior to bringing the patient in for their first study visit.
2. The eligible patient must meet the data requirements as specified in the protocol, i.e., baseline data collected within 7 days prior to treatment with ILUVIEN and additional data subsequently collected approximately every 6 months thereafter until enrolment into the study.
3. The eligible patient must be enrolled at least one year prior to the planned end of the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with vision impairment associated with chronic diabetic macular oedema considered insufficiently responsive to available therapies that were selected to be treated with an intravitreal implant of ILUVIEN.
Sampling Method: Non-Probability Sample
Enrollment: 559 (Actual)
Dates: Start 2013-12; Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events. | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Atlanta, Georgia, United States

REFERENCES:
- [Result] Chakravarthy U, Taylor SR, Koch FHJ, Castro de Sousa JP, Bailey C; ILUVIEN Registry Safety Study (IRISS) Investigators Group. Changes in intraocular pressure after intravitreal fluocinolone acetonide (ILUVIEN): real-world experience in three European countries. Br J Ophthalmol. 2019 Aug;103(8):1072-1077. doi: 10.1136/bjophthalmol-2018-312284. Epub 2018 Sep 21. PMID 30242062
- See also: Changes in intraocular pressure after intravitreal fluocinolone acetonide (ILUVIEN): real-world experience in three European countries — http://dx.doi.org/10.1136/bjophthalmol-2018-312284